CLINICAL TRIAL: NCT06190912
Title: A Single-Arm, Single-Site, Single-Dose Phase 1 Study Assessing the Safety of Bryostatin in the Treatment of Patients With Multiple Sclerosis
Brief Title: Safety of Bryostatin in Patients With MS
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Fox (Other)
Collaborators: Synaptogenix, Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Robert Fox, Vice Chair for Research, Neurological Institute, Staff Neurologist, Cleveland Clinic Mellen Center for MS Treatment and Research, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-099
Record Dates: First submitted 2023-12-11; First posted 2024-01-05 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — bryostatin 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bryostatin 1 (Experimental): Participants in this arm will receive treatment with Bryostatin 1
  Interventions: Drug: Bryostatin 1

INTERVENTIONS:
Drug: Bryostatin 1 — Eligible participants will be treated with bryostatin over a 26-week period. Doses 1, 2, 8, and 9 of the study drug will be a loading dose 20% higher (i.e., 24 µg) than the assigned fixed dose and will be administered one week apart. Otherwise, the assigned fixed dose is 20 µg. Drug is administered intravenously (IV) by continuous infusion over 45(±5) minutes. Participants are scheduled to receive 14 doses over 26 weeks.

SUMMARY:
This is a single-site, single-arm, single-dose, Phase 1 study of the safety of bryostatin in participants with multiple sclerosis (MS) receiving any disease modifying therapy (DMT).

DETAILED DESCRIPTION:
The study is 42 weeks in duration, including safety and exploratory outcomes evaluation at 30 days after the last full assessment (Week 28) and long-term follow-up at 12 weeks after the last full assessment (Week 40). Participants will receive a total of 14 doses over 26 weeks.

Eligible participants will be treated with bryostatin over a 26-week period. Doses 1, 2, 8, and 9 of the study drug will be a loading dose 20% higher (i.e., 24 µg) than the assigned fixed dose and will be administered one week apart. Otherwise, the assigned fixed dose is 20 µg. Drug is administered intravenously (IV) by continuous infusion over 45 (±5) minutes. Participants are scheduled to receive 14 doses over 26 weeks.

ELIGIBILITY:
Inclusion

1. Written informed consent signed by participant
2. English-speaking
3. Hospital Anxiety and Depression Scale <11
4. Male and female participants, 18-65 years of age inclusive
5. Established diagnosis of MS, as defined by the 2017 revision of McDonald Diagnostic Criteria (any form of MS). A diagnosis of MS must be confirmed at the time of the screening visit.
6. Processing Speed Test (PST) z-score between -1.0 and -2.5
7. EDSS between 0.0 and 7.0, inclusive.
8. Adequate vision and motor function to participate in assessment procedures
9. Participants must be off of a DMT or on a stable dose of a DMT for at least 1 year prior to entry into the study, and the dose should not change during the study unless a change is required by a clinically significant change in the participant's status.
10. Females participating in the study must meet one the following criteria:

    1. Surgically sterilized (e.g., hysterectomy, bilateral oophorectomy or tubal ligation) for at least 6 months or postmenopausal (postmenopausal females must have no menstrual bleeding for at least 1 year) or
    2. If not postmenopausal, agree to use a double method of contraception, one of which is a barrier method (e.g., intrauterine device plus condom, spermicidal gel plus condom) 30 days prior to dosing until 30 days after last dose and have negative human chorionic gonadotropin (β-hCG) test for pregnancy at screening. Contraception methods resulting in an overall failure rate of <1 % per year are required for women of childbearing potential.
11. Males who have not had a vasectomy must use appropriate contraception methods (barrier or abstinence) from 30 days prior to dosing until 30 days after last dose
12. Participants should be in reasonably good health over the last 6 months and any chronic disease should be stable.

Exclusion

1. Evidence of significant CNS vascular disease on previous neuroimaging, including but not limited to cortical stroke, multiple infarcts, localized single infarcts in the thalamus, angular gyrus, multiple lacunar infarcts, or extensive white matter injury
2. Clinically significant neurologic disease or condition other than MS, such as cerebral tumor, chronic subdural fluid collections, Huntington's Disease, Parkinson's Disease, normal pressure hydrocephalus, or any other diagnosis that could interfere with assessment of safety and efficacy
3. Previous history of seizures or seizure disorders.
4. Evidence of clinically significant unstable cardiovascular, pulmonary, renal, hepatic, gastrointestinal, neurologic, or metabolic disease within the 6 months prior to enrollment. If there is a history of cancer, the participant should be clear of cancer for at least 2 years prior to screening. More recent history of basal cell or squamous cell carcinoma and melanoma in situ (Stage 0) may be acceptable after review by the Medical Monitor.
5. Estimated Glomerular Filtration Rate (eGFR) of <45ml/min
6. Poorly controlled diabetes (at the discretion of the Principal Investigator)
7. Use of vitamin E > 400 International Units (IU) per day within 14 days prior to screening
8. Use of valproic acid and/or lithium within 14 days prior to screening
9. Use of carbamazepine within 7 days prior to screening
10. Use of teriflunomide within 90 days prior to screening
11. Use of dalfampridine within 7 days of screening
12. Current use of acetaminophen, ciprofloxacin, and/or trimethoprim/sulfamethoxazole
13. Use of any potent or moderate inhibitor or inducer of CYP3A4, CYP2C8, or CYP2C9. Concomitant medicines will be examined on a case-by-case basis against the Flockhart Table by study investigator, and if needed, the Medical Monitor, to determine allowability
14. Current use of St. John's Wort, within 2 weeks prior to screening
15. Consumption of grapefruit juice from screening until end of study
16. At the discretion of the PI, any medical or psychiatric condition that is unstable or may require the initiation of additional medication or surgical intervention during the course of the study
17. Any screening laboratory values outside the laboratory reference ranges that are deemed clinically significant by the PI
18. Use of an investigational drug within 30 days prior to screening
19. Suicidality defined as active suicidal thoughts during the 6 months prior to screening or at Baseline [SBQ-R], or history of suicide attempt in previous 2 years, or at serious suicide risk in study neurologist or PI's judgment
20. Major psychiatric illness such as currently uncontrolled major depression according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition4, current or past diagnosis of bipolar disorder, schizophrenia, or any other psychiatric disorder that might interfere with the assessments of safety or efficacy at the discretion of the PI
21. Diagnosis of alcohol or drug abuse within the last 2 years
22. History of prolonged QT or prolonged QT on screening ECG [QT correction with Bazett formula (QTcB) or QT correction by Fridericia (QTcF)>499 per central reader]5
23. Acute or poorly controlled medical illness: blood pressure >180 mmHg systolic or 100 mmHg diastolic; myocardial infarction within 6 months; uncompensated congestive heart failure [New York Heart Association (NYHA) Class III or IV]
24. Known to be seropositive for Hepatitis B or C, unless successful curative treatment for Hepatitis C (e.g., Harvoni) has been received, and there is documentation that there is no Hepatitis B/C virus detected 3 months after completion of treatment
25. Known to be seropositive for human immunodeficiency virus (HIV)
26. Pregnancy or breastfeeding during the study. A β-hCG serum pregnancy test will be performed at Screening for female patients of child-bearing potential.
27. Aspartate Amino Transferase (AST) or Alanine Aminotransferase (ALT) >3x upper limit of normal (ULN) and total bilirubin >2x ULN or International Normalized Ratio (INR) >1.5
28. History of significant bleeding disorders.
29. Moderate baseline thrombocytopenia (platelets <100K/uL).
30. Elevated INR (>2.0).
31. Prior exposure to bryostatin, or known sensitivity to bryostatin or any ingredient in the study drug
32. Any other concurrent medical condition, which in the opinion of the PI makes the participant unsuitable for the clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Over 40 weeks
  Frequency of Adverse Events [Treatment Emergent AEs (TEAEs), Serious Adverse Events (SAEs), and Suspected Unexpected Serious Adverse Reactions (SUSARS)]
Study Medication Discontinuation | Over 40 weeks
  Frequency of study medication discontinuation and reason thereof
CNS inflammatory effects | Over 40 weeks
  Potential CNS inflammatory effects as captured by clinical monitoring and MRI

OTHER OUTCOMES:
Exploratory outcome: MRI Biomarkers (lesion volume) | Changes from baseline to Week 11, Week 28, and Week 40
  Lesion volume
Exploratory outcome: MRI Biomarkers (BPF) | Changes from baseline to Week 11, Week 28, and Week 40
  Brain parenchymal fraction
Exploratory outcome: MRI Biomarkers (default mode network) | Changes from baseline to Week 11, Week 28, and Week 40
  Default mode network
Exploratory outcome: MRI Biomarkers (microstructural complexity of dendrites and axons) | Changes from baseline to Week 11, Week 28, and Week 40
  Diffusion MRI measures of tissue integrity
Exploratory outcome: MRI Biomarkers (anatomical connectivity of transcallosal motor pathway) | Changes from baseline to Week 11, Week 28, and Week 40
  Anatomical connectivity of transcallosal motor pathway
Exploratory outcome: MRI Biomarkers (MWF) | Changes from baseline to Week 11, Week 28, and Week 40
  Myelin water fraction
Exploratory outcome: MRI Biomarkers (measure of myelination) | Changes from baseline to Week 11, Week 28, and Week 40
  Magnetization transfer ratio
Exploratory outcome: MRI Biomarkers (measure of myelination) | Changes from baseline to Week 11, Week 28, and Week 40
  Quantitative T2*
Exploratory outcome: MRI Biomarkers (measure of myelination) | Changes from baseline to Week 11, Week 28, and Week 40
  Quantitative susceptibility mapping
Exploratory outcome: MRI Biomarkers (GMA) | Changes from baseline to Week 11, Week 28, and Week 40
  Grey matter atrophy
Exploratory outcome: MRI Biomarkers (GMF) | Changes from baseline to Week 11, Week 28, and Week 40
  Grey matter fraction
Exploratory outcome: MRI Biomarkers (WMF) | Changes from baseline to Week 11, Week 28, and Week 40
  White matter fraction
Exploratory outcome: MRI Biomarkers (CA) | Changes from baseline to Week 11, Week 28, and Week 40
  Cortical atrophy
Exploratory Outcome: MoCA | Changes from baseline to Week 11, Week 28, and Week 40
  Montreal Cognitive Assessment test
Exploratory Outcome: EDSS | Changes from baseline to Week 11, Week 28, and Week 40
  Expanded Disability Status Scale
Exploratory Outcomes: MS Performance Test Domains (Lower Extremity) | Changes from baseline to Week 11, Week 28, and Week 40
  Walking Speed Test (WST)
Exploratory Outcomes: MS Performance Test Domains (Upper Extremity) | Changes from baseline to Week 11, Week 28, and Week 40
  Manual dexterity test (MDT)
Exploratory Outcomes: MS Performance Test Domains (Cognition) | Changes from baseline to Week 11, Week 28, and Week 40
  Processing speed test (PST)
Exploratory Outcomes: Quality of life (NEURO-QoL) | Changes from baseline to Week 11, Week 28, and Week 40
  Quality of Life in Neurological Disorders (NEURO-QoL)
Exploratory Outcomes: CVLT3 | Change from baseline to Week 28 and Week 40
  California Verbal Learning Test 3rd Edition (CVLT3)
Exploratory Outcomes: BVMT-R | Change from baseline to Week 28 and Week 40
  Brief Visuospatial Memory Test - Revised (BVMT-R)
Exploratory Outcomes: JOLO | Change from baseline to Week 28 and Week 40
  Judgement of Line Orientation (JOLO)
Exploratory Outcomes: BNT | Change from baseline to Week 28 and Week 40
  Boston Naming Test (BNT)
Exploratory Outcomes: D-KEFS (Sorting) | Change from baseline to Week 28 and Week 40
  Delis-Kaplan Executive Function System (D-KEFS) Sorting Test
Exploratory Outcomes: COWAT | Change from baseline over 40 weeks
  Controlled Oral Word Association Test

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Fox, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No